CLINICAL TRIAL: NCT01670032
Title: A Multicenter, Double Blind, Randomized, Vehicle Controlled Study to Evaluate the Efficacy and Safety of Two Dose Regimens of CD 07223 1.5% Topical Gel in Impetigo
Brief Title: Vehicle Controlled Efficacy and Safety Study of Two Dose Regimens of CD07223 1.5% Topical Gel in Impetigo
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NovaBay Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.06. SPR. 18216
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Impetigo
MeSH Terms: conditions — Impetigo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CD07223 1.5 % Topical Gel BID (Experimental): Drug: 1.5% CD07223 Topical Gel applied BID for 7 days
  Interventions: Drug: Experimental: CD07223 1.5 % Topical Gel BID
- CD07223 1.5% Topical Gel TID (Experimental): Drug: 1.5% CD07223 Topical Gel applied TID for 7 days
  Interventions: Drug: Experimental: CD07223 1.5% Topical Gel TID
- CD07223 vehicle gel BID (Placebo Comparator): Drug: CD07223 Vehicle Topical Gel applied BID for 7 days
  Interventions: Drug: Placebo Comparator: CD07223 vehicle gel BID
- CD07223 vehicle gel TID (Placebo Comparator): Drug: CD07223 Vehicle Topical Gel applied TID for 7 days
  Interventions: Drug: Placebo Comparator: CD07223 vehicle gel TID

INTERVENTIONS:
Drug: Experimental: CD07223 1.5 % Topical Gel BID — Eligible subjects are to apply study medication twice a day (BID) for seven days. All lesions will be treated with study medication. Scheduled study visits will occur at Day 1, Day 3, Day 8 and Day 15
  Arms: CD07223 1.5 % Topical Gel BID
Drug: Experimental: CD07223 1.5% Topical Gel TID — Eligible subjects are to apply study medication three times a day (TID) for seven days. All lesions will be treated with study medication. Scheduled study visits will occur at Day 1, Day 3, Day 8 and Day 15
  Arms: CD07223 1.5% Topical Gel TID
Drug: Placebo Comparator: CD07223 vehicle gel BID — Eligible subjects are to apply study medication twice a day (BID) for seven days. All lesions will be treated with study medication. Scheduled study visits will occur at Day 1, Day 3, Day 8 and Day 15
  Arms: CD07223 vehicle gel BID
Drug: Placebo Comparator: CD07223 vehicle gel TID — Eligible subjects are to apply study medication three times a day (TID) for seven days. All lesions will be treated with study medication. Scheduled study visits will occur at Day 1, Day 3, Day 8 and Day 15
  Arms: CD07223 vehicle gel TID

SUMMARY:
This study will be a multicenter, randomized, vehicle controlled, parallel, group, double blind study. Eligible subjects with a clinical diagnosis of impetigo will be randomized to one of four treatment groups: 1.5% CD07223 Topical Gel applied BID; 1.5% CD07223 Topical Gel applied TID; Vehicle Topical Gel applied BID;Vehicle Topical Gel applied TID. All treatments will be administered for 7 days. Disease activity for the Target Lesion will be evaluated using the Skin Infection Rating Scale (SIRS) Score.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 2 years of age or older
* Clinical diagnosis of primary impetigo (bullous or non bullous)
* Minimum diameter of Target Lesion to be one centimeter measured either as length or width.
* Presence of at least one and no more than ten lesions per subject at the time of screening
* The infected lesions' total area (as determined by the Investigator) must be less than 100 cm2 in total area for subjects 18 years of age or older, or up to a maximum of 2% total body surface area for subjects younger than 18 years of age.
* Skin Infection Rating Scale (SIRS) total score of the Target Lesion of at least 4

Exclusion Criteria:

* Presence of other active skin diseases at or near the Target Lesion area to be treated
* A subject whose disease is so widespread or severe that, in the opinion of the investigator, oral antibiotic treatment is needed
* Signs and symptoms of another current infection requiring antibiotic treatment
* Tympanic temperature at Screening/Baseline exceeding 38 degrees Celsius (100.4 degrees Fahrenheit) in a pediatric subject or 37.8 degrees Celsius (100 degrees Fahrenheit) in an adult subject
* History of Hepatitis B or C, HIV/ AIDS, or other immunodeficiency disease
* Concurrent or recent scabies infection or lice infestation (pediculosis) of the scalp
* Use of systemic antibiotics or systemic steroids within 14 days prior to study entry. A history of three or more courses of systemic antibiotics within the 3 month period immediately prior to screening will also be considered exclusionary
* Use of topical antibiotics, topical antibacterials, topical antifungals or topical steroids within 14 days prior to study entry on any skin lesion (as deemed significant by the Investigator by virtue of the lesion's nature and/or position to impact on the effectiveness of the study drug)
* Participation in any other clinical study or use of any investigational drugs or investigational device within 30 days prior to enrollment
* Presence of secondarily infected traumatic lesions (e.g. surgical wounds, animal/insect bites, burns, lacerations and abrasions).
* Another family member in same household currently enrolled in this study or another family member in the same household with active impetigo

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Clinical Success at Follow up (Day 15) in the intent-to-treat (ITTC) population | 2 weeks
  Clinical Success is defined by the SIRS score of the Target Lesion

CONTACTS AND LOCATIONS:
Locations (13):
- United States (7):
  - SRCR, Inc, Bell Gardens, California
  - Skin Care research Inc, Boca Raton, Florida
  - Eastern Research, Inc, Hialeah, Florida
  - Cyn3rgy Research, Gresham, Oregon
  - Cheraw Pediatrics, P.A., Cheraw, South Carolina
  - Integrity Clinical Research, Inc, Milan, Tennessee
  - Sealy Urgent Care Center, Sealy, Texas
- South Africa (6):
  - Langeberg Clinical Trials, Kraaifontein, Cape Town
  - Newtown Clinical Research, Johannesburg, Gauteng
  - Phelang Research Center, Pretoria, Gauteng
  - Setshaba Research Center, Soshanguve, Gauteng
  - Welkom Clinical Trial Center, Welkom, Gauteng
  - Synopsis Research, Rondebosch, Western Cape